CLINICAL TRIAL: NCT02116946
Title: Intratendinous Injections of Platelet Rich Plasma With or Without Leukocyte Enrichment for Patellar Tendinopathy: a Randomized Controlled Trial
Brief Title: Plasma Injections Plus Exercise for Patellar Tendinopathy
Acronym: PHS
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: 79% participant retention after 1 year
Sponsor: University of British Columbia (Other)
Collaborators: American Orthopaedic Society for Sports Medicine (Other); University of Washington (Other); Rizzoli Orthopaedic Institute (Unknown); Norwegian Olympic Sports Center (Unknown); University of Oslo (Other); Steadman Clinic (Unknown)
Responsible Party: Principal Investigator, Alexander Scott, Principal Investigator, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: H13-00254
Record Dates: First submitted 2014-04-09; First posted 2014-04-17 (Estimated); Last update posted 2018-12-21 (Actual); Status verified 2018-12

CONDITIONS: Patellar Tendinopathy
MeSH Terms: interventions — Poverty; Sodium Chloride; Exercise

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Leukocyte-rich Platelet Rish Plasma + exercise (Experimental): Leukocyte-rich PRP injection and a 12 week exercise program.
  Interventions: Biological: Platelet Rich Plasma (PRP)
- Leukocyte-poor Platelet Rich Plasma + exercise (Experimental): Leukocyte-poor PRP injection and a 12 week exercise program.
  Interventions: Biological: Platelet Rich Plasma (PRP)
- Saline + exercise (Placebo Comparator): Saline injection and a 12 week exercise program.
  Interventions: Other: Saline + exercise

INTERVENTIONS:
Biological: Platelet Rich Plasma (PRP) — Injection of Leukocyte-rich or Leukocyte-poor Platelet Rich Plasma prepared by the Angel cPRP System along with a 12 week exercise program for treatment of patients with patellar tendinopathy.
  Other Names: The device Angel cPRP System will be used to make (Leukocyte-rich or -poor) PRP injections
  Arms: Leukocyte-poor Platelet Rich Plasma + exercise; Leukocyte-rich Platelet Rish Plasma + exercise
Other: Saline + exercise — Peritendinous saline injection plus 12 week exercise program.
  Arms: Saline + exercise

SUMMARY:
This is a randomized controlled clinical trial to investigate the effectiveness, safety and tolerability of platelet-rich plasma (PRP) injections for treatment of patellar tendinopathy in adults 18-50 years of age. Subjects will be randomly assigned to three parallel treatment groups:

1. Leukocyte-rich PRP injection + exercise
2. Leukocyte-poor PRP injection + exercise
3. Saline injection + exercise (control) Primary endpoints are (1) the number (rate) and severity of adverse events as reported by both patients and study physicians during the first 12 weeks after initiation of treatment, (2) patient-rated tolerability of treatment; (3) the change in function (VISA score) and treatment success (global improvement scale) over six months of a post-injection exercise protocol.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥ 18 and ≤ 50 years of age at Enrollment Visit
* Documentation of a clinical diagnosis of patellar tendinopathy, grade-IIIB Blazina stage, confirmed on ultrasound
* Previously tried an exercise program of at least six weeks duration
* Fluent in official language of study site
* Written informed consent obtained from subject
* Normal values on screening laboratory panels (CBC, PT, PTT, INR, serum creatine, ALT, ALP, AST, bilirubin, albumin)

Exclusion Criteria:

* For women of child-bearing potential, positive pregnancy test at enrollment visit
* Major surgery in the past three months
* Surgery on the symptomatic knee
* Bleeding disorder
* Systemic inflammatory disease
* Arthritis or degenerative knee condition
* Recent fluoroquinolone use
* Subjects who have any requirement for the use of systemic steroids or immunosuppressants
* Subjects who are known to be HIV positive
* Uncooperative patient, or patients who are incapable of following directions or who are predictably unwilling to return for follow-up examinations
* Presence of a condition or abnormality that in the opinion of the Investigator would compromise the safety of the patient or the quality of the data

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2014-03; Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Clinical Efficacy | 2 years
  Number and frequency of adverse events will be assessed/reported weekly for the first 12 weeks and at the 6 month visit.

SECONDARY OUTCOMES:
Change in function over time measured by VISA Score | 2 years
  To compare change in function (VISA score) between participants randomized to the three treatment groups over six months, 1 year, and 2 years of a post-injection exercise protocol.
Comparison of treatment success measured by Likert Global Improvement Scale | 2 years
  To compare change in treatment success (Likert global improvement scale) between participants randomized to the three treatment groups over six months, 1 year, and 2 years of a post-injection exercise protocol.
Change in activity levels over time measured by Tegner Activity Score | 2 years
  To compare change in activity levels (Tegner Activity Score) between participants randomized to the three groups over six months, 1 year, and 2 years of an exercise protocol.
Change in activity-related pain over time measured by Pain Numeric Rating Scale | 2 years
  To compare change in activity-related pain (Pain Numeric Rating Scale) between participants randomized to the three groups over six months, 1 year, and 2 years of an exercise protocol.

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Scott, PhD, Principal Investigator — University of British Columbia
Locations (5):
- United States (2):
  - The Steadman Clinic, Vail, Colorado
  - University of Washington, Seattle, Washington
- University of Britich Columbia, Vancouver, British Columbia, Canada
- Rizzoli Orthopaedic Institute, Bologna, Italy
- Oslo Sports Trauma Research Center, Oslo, Norway

REFERENCES:
- [Background] Lian OB, Engebretsen L, Bahr R. Prevalence of jumper's knee among elite athletes from different sports: a cross-sectional study. Am J Sports Med. 2005 Apr;33(4):561-7. doi: 10.1177/0363546504270454. Epub 2005 Feb 8. PMID 15722279
- [Background] Ferretti A. Epidemiology of jumper's knee. Sports Med. 1986 Jul-Aug;3(4):289-95. doi: 10.2165/00007256-198603040-00005. PMID 3738327
- [Background] Lian O, Engebretsen L, Ovrebo RV, Bahr R. Characteristics of the leg extensors in male volleyball players with jumper's knee. Am J Sports Med. 1996 May-Jun;24(3):380-5. doi: 10.1177/036354659602400322. PMID 8734892
- [Background] Engebretsen L, Steffen K, Alsousou J, Anitua E, Bachl N, Devilee R, Everts P, Hamilton B, Huard J, Jenoure P, Kelberine F, Kon E, Maffulli N, Matheson G, Mei-Dan O, Menetrey J, Philippon M, Randelli P, Schamasch P, Schwellnus M, Vernec A, Verrall G. IOC consensus paper on the use of platelet-rich plasma in sports medicine. Br J Sports Med. 2010 Dec;44(15):1072-81. doi: 10.1136/bjsm.2010.079822. No abstract available. PMID 21106774
- [Background] Scott, A, KM Khan, J Cook, and V Duronio, Human tendon overuse pathology: histopathologic and biochemical findings, in Tendinopathy in Athletes, S.L. Woo, S.P. Arnoczky, and P. Renstrom, Editors. 2007, Blackwell Publishing Ltd: Malden, Massachusetts. p. 69-84.
- [Background] Kongsgaard M, Qvortrup K, Larsen J, Aagaard P, Doessing S, Hansen P, Kjaer M, Magnusson SP. Fibril morphology and tendon mechanical properties in patellar tendinopathy: effects of heavy slow resistance training. Am J Sports Med. 2010 Apr;38(4):749-56. doi: 10.1177/0363546509350915. Epub 2010 Feb 12. PMID 20154324
- [Background] Larsson ME, Kall I, Nilsson-Helander K. Treatment of patellar tendinopathy--a systematic review of randomized controlled trials. Knee Surg Sports Traumatol Arthrosc. 2012 Aug;20(8):1632-46. doi: 10.1007/s00167-011-1825-1. Epub 2011 Dec 21. PMID 22186923
- [Background] Bahr R, Fossan B, Loken S, Engebretsen L. Surgical treatment compared with eccentric training for patellar tendinopathy (Jumper's Knee). A randomized, controlled trial. J Bone Joint Surg Am. 2006 Aug;88(8):1689-98. doi: 10.2106/JBJS.E.01181. PMID 16882889
- [Background] Warden SJ, Metcalf BR, Kiss ZS, Cook JL, Purdam CR, Bennell KL, Crossley KM. Low-intensity pulsed ultrasound for chronic patellar tendinopathy: a randomized, double-blind, placebo-controlled trial. Rheumatology (Oxford). 2008 Apr;47(4):467-71. doi: 10.1093/rheumatology/kem384. Epub 2008 Feb 12. PMID 18270224
- [Background] Kongsgaard M, Kovanen V, Aagaard P, Doessing S, Hansen P, Laursen AH, Kaldau NC, Kjaer M, Magnusson SP. Corticosteroid injections, eccentric decline squat training and heavy slow resistance training in patellar tendinopathy. Scand J Med Sci Sports. 2009 Dec;19(6):790-802. doi: 10.1111/j.1600-0838.2009.00949.x. Epub 2009 May 28. PMID 19793213
- [Background] Rees JD, Maffulli N, Cook J. Management of tendinopathy. Am J Sports Med. 2009 Sep;37(9):1855-67. doi: 10.1177/0363546508324283. Epub 2009 Feb 2. PMID 19188560
- [Background] van Ark M, Zwerver J, van den Akker-Scheek I. Injection treatments for patellar tendinopathy. Br J Sports Med. 2011 Oct;45(13):1068-76. doi: 10.1136/bjsm.2010.078824. Epub 2011 May 3. PMID 21543346
- [Background] Filardo G, Kon E, Della Villa S, Vincentelli F, Fornasari PM, Marcacci M. Use of platelet-rich plasma for the treatment of refractory jumper's knee. Int Orthop. 2010 Aug;34(6):909-15. doi: 10.1007/s00264-009-0845-7. Epub 2009 Jul 31. PMID 19641918
- [Background] Kon E, Filardo G, Delcogliano M, Presti ML, Russo A, Bondi A, Di Martino A, Cenacchi A, Fornasari PM, Marcacci M. Platelet-rich plasma: new clinical application: a pilot study for treatment of jumper's knee. Injury. 2009 Jun;40(6):598-603. doi: 10.1016/j.injury.2008.11.026. Epub 2009 Apr 19. PMID 19380129
- [Background] Banfi G, Corsi MM, Volpi P. Could platelet rich plasma have effects on systemic circulating growth factors and cytokine release in orthopaedic applications? Br J Sports Med. 2006 Oct;40(10):816. doi: 10.1136/bjsm.2006.029934. Epub 2006 Aug 18. No abstract available. PMID 16920768
- [Background] Sheth U, Simunovic N, Klein G, Fu F, Einhorn TA, Schemitsch E, Ayeni OR, Bhandari M. Efficacy of autologous platelet-rich plasma use for orthopaedic indications: a meta-analysis. J Bone Joint Surg Am. 2012 Feb 15;94(4):298-307. doi: 10.2106/JBJS.K.00154. PMID 22241606
- [Background] Thanasas C, Papadimitriou G, Charalambidis C, Paraskevopoulos I, Papanikolaou A. Platelet-rich plasma versus autologous whole blood for the treatment of chronic lateral elbow epicondylitis: a randomized controlled clinical trial. Am J Sports Med. 2011 Oct;39(10):2130-4. doi: 10.1177/0363546511417113. Epub 2011 Aug 2. PMID 21813443
- [Background] Castillo TN, Pouliot MA, Kim HJ, Dragoo JL. Comparison of growth factor and platelet concentration from commercial platelet-rich plasma separation systems. Am J Sports Med. 2011 Feb;39(2):266-71. doi: 10.1177/0363546510387517. Epub 2010 Nov 4. PMID 21051428
- [Background] Dragoo JL, Braun HJ, Durham JL, Ridley BA, Odegaard JI, Luong R, Arnoczky SP. Comparison of the acute inflammatory response of two commercial platelet-rich plasma systems in healthy rabbit tendons. Am J Sports Med. 2012 Jun;40(6):1274-81. doi: 10.1177/0363546512442334. Epub 2012 Apr 10. PMID 22495144
- [Background] Dworkin RH, Turk DC, Farrar JT, Haythornthwaite JA, Jensen MP, Katz NP, Kerns RD, Stucki G, Allen RR, Bellamy N, Carr DB, Chandler J, Cowan P, Dionne R, Galer BS, Hertz S, Jadad AR, Kramer LD, Manning DC, Martin S, McCormick CG, McDermott MP, McGrath P, Quessy S, Rappaport BA, Robbins W, Robinson JP, Rothman M, Royal MA, Simon L, Stauffer JW, Stein W, Tollett J, Wernicke J, Witter J; IMMPACT. Core outcome measures for chronic pain clinical trials: IMMPACT recommendations. Pain. 2005 Jan;113(1-2):9-19. doi: 10.1016/j.pain.2004.09.012. No abstract available. PMID 15621359
- [Background] Briggs KK, Steadman JR, Hay CJ, Hines SL. Lysholm score and Tegner activity level in individuals with normal knees. Am J Sports Med. 2009 May;37(5):898-901. doi: 10.1177/0363546508330149. Epub 2009 Mar 23. PMID 19307332
- [Derived] Scott A, LaPrade RF, Harmon KG, Filardo G, Kon E, Della Villa S, Bahr R, Moksnes H, Torgalsen T, Lee J, Dragoo JL, Engebretsen L. Platelet-Rich Plasma for Patellar Tendinopathy: A Randomized Controlled Trial of Leukocyte-Rich PRP or Leukocyte-Poor PRP Versus Saline. Am J Sports Med. 2019 Jun;47(7):1654-1661. doi: 10.1177/0363546519837954. Epub 2019 Apr 30. PMID 31038979